CLINICAL TRIAL: NCT05780567
Title: Randomized, Double-blind, Parallel-controlled Phase III Trial to Evaluate the Efficacy and Safety of TQB3616 Combined With Endocrine Therapy Versus Placebo Combined With Endocrine Therapy in Hormone Receptors (HR)-Positive and Human Epidermal GrowthFactor Receptor-2 (HER2) -Negative Breast Cancer Adjuvant Therapy
Brief Title: Clinical Study on Adjuvant Therapy of TQB3616 Combined With Endocrine Therapy Compared With Placebo Combined With Endocrine Therapy in Patients With Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQB3616-III-03
Record Dates: First submitted 2023-03-10; First posted 2023-03-22 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Anastrozole; Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB3616 capsules combined with endocrine (Experimental): The dose of TQB3616 capsules is 180mg, taken orally when fasting, once a day for 28 consecutive days as one treatment cycle.
  The dose of Letrozole is 2.5mg, taken orally, once a day for 28 consecutive days as one treatment cycle.
  The dose of Anastrozole is 1mg, taken orally, once a day for 28 consecutive days as one treatment cycle.
  The dose of Tamoxifen is 10mg, taken orally, twice a day for 28 consecutive days as one treatment cycle.
  Interventions: Drug: TQB3616 capsules, Letrozole, Anastrozole, Tamoxifen
- placebo combined with endocrine (Placebo Comparator): The dose of placebo is 180mg, taken orally when fasting, once a day for 28 consecutive days as one treatment cycle.
  The dose of Letrozole is 2.5mg, taken orally, once a day for 28 consecutive days as one treatment cycle.
  The dose of Anastrozole is 1mg, taken orally, once a day for 28 consecutive days as one treatment cycle.
  The dose of Tamoxifen is 10mg, taken orally, twice a day for 28 consecutive days as one treatment cycle.
  Interventions: Drug: Placebo capsules, Letrozole, Anastrozole, Tamoxifen

INTERVENTIONS:
Drug: TQB3616 capsules, Letrozole, Anastrozole, Tamoxifen — TQB3616 is a novel Cyclin-dependent kinase (CDK) 4/6 inhibitor and currently being used in the treatment of a variety of malignant solid tumors.
  Letrozole combined with Anastrozole and Tamoxifen is an endocrine therapy that involves adding, blocking, or removing hormones. It can be used for conditions that affect hormone levels, such as breast cancer.
  Arms: TQB3616 capsules combined with endocrine
Drug: Placebo capsules, Letrozole, Anastrozole, Tamoxifen — Letrozole combined with Anastrozole and Tamoxifen is an endocrine therapy that involves adding, blocking, or removing hormones. It can be used for conditions that affect hormone levels, such as breast cancer.
  Arms: placebo combined with endocrine

SUMMARY:
This is a Phase III, randomized, double-blind, parallel, multi-center trail to evaluate the efficacy and safety of TQB3616 capsule combined with endocrine compared to placebo compared with endocrine in HR-positive and HER2-negative breast cancer adjuvant therapy. Approximately 1946 female subjects will be randomized to either TQB3616 combined with endocrine group or TQB3616-matching placebo combined endocrine group. Randomization will follow a 2:1 ratio, 1297 subjects in experimental group and 649 in the the Placebo Comparator group.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined the study and signed the informed consent, with good compliance.
* Age: 18-75 years old (upon signing the informed consent); Eastern Cooperative Oncology Group Performance Status (PS) score: 0~1;
* Surgical treatment of radical mastectomy;
* Pathological examination confirmed HR positive and HER2 negative invasive breast cancer;
* The major organs are functioning well, meeting the following criteria：

  1. Blood biochemical tests should meet the following criteria (no corrective therapy has been used within 7 days prior to screening)：

     1. Hemoglobin (HB) ≥90 g/L；
     2. Neutrophil absolute value (NEUT) ≥ 1.5×109/L；
     3. Platelet count (PLT) ≥ 100 ×109/L；
  2. Blood biochemical tests should meet the following criteria (no corrective therapy has been used within 7 days prior to screening)：

     1. Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN)；
     2. Alanine transferase (ALT) and aspartate transferase (AST) ≤ 1.5×ULN；
     3. Serum creatinine (Cr) ≤ 1.5×ULN, or creatinine clearance (Ccr) ≥ 60 ml/min；
  3. Blood clotting tests must meet the following criteria (no anticoagulant therapy)：

     1. Prothrombin time (PT) ≤ 1.5×ULN;
     2. Activated partial thromboplastin time (APTT) ≤ 1.5×ULN;
     3. International Normalized ratio (INR) ≤ 1.5×ULN.
  4. Left ventricular ejection fraction (LVEF) ≥50%.

Exclusion Criteria:

* Complicated diseases and medical history:

  1. Has had other malignant tumors within 5 years or currently has other malignant tumors;
  2. Have a variety of factors that affect oral medication (such as inability to swallow);
  3. Current history of serious lung disease such as interstitial pneumonia；
  4. Severe infections common terminology criteria for adverse events (≥CTCAE (common terminology criteria for adverse events) 2 grade) that were active or uncontrolled before the study treatment started (Except hair loss and hemoglobin)；
* Known allergy to aromatase inhibitors, tamoxifen, TQB3616/ placebo, or any excipients;
* There was a history of live attenuated vaccine vaccination within 28 days prior to randomization or live attenuated vaccine vaccination was planned during the study period;
* Participated in clinical trials of other antitumor agents within 4 weeks prior to randomization；
* The presence of other serious physical or mental illnesses or abnormalities in laboratory tests that may increase the risk of study participation or interfere with the study results, as well as subjects who are deemed unsuitable for study participation for other reasons by the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1946 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease-Free Survival (IDFS) | Baseline up to 60 months
  The time from the date of randomization to the first occurrence of the following events, including ipsilateral or contralateral recurrence of invasive breast cancer, regional or distant recurrence of invasive breast cancer, secondary primary malignancy outside the breast, and death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | Baseline up to 60 months
  The time from first administration to death of any cause.
Disease Relapse Free Survival (DRFS) | Baseline up to 60 months
  The time from the date of randomization to the first occurrence of distant recurrence or death from any cause.
Incidence of adverse events | Baseline up to 60 months
  Incidence of adverse events assessed according to the common terminology criteria for adverse events (CTCAE).
Severity of adverse events | Baseline up to 60 months
  Severity of adverse events assessed according to the common terminology criteria for adverse events (CTCAE).
Incidence of abnormal laboratory test values | Baseline up to 60 months
  Incidence of abnormal laboratory test values assessed according to the common terminology criteria for adverse events (CTCAE).
Severity of abnormal laboratory test values | Baseline up to 60 months
  Severity of abnormal laboratory test values assessed according to the common terminology criteria for adverse events (CTCAE).
Incidence of serious adverse events | Baseline up to 60 months
  Incidence of serious adverse events assessed according to the common terminology criteria for adverse events (CTCAE).
Severity of serious adverse events | Baseline up to 60 months
  Severity of serious adverse events assessed according to the common terminology criteria for adverse events (CTCAE).

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Suining Central Hospital, Suining, Sichuan